CLINICAL TRIAL: NCT07181226
Title: High-Frequency vs. Theta-Burst TMS in Depression: Head-to-Head Double-Blind Randomized Trial With Six-week Follow-up
Brief Title: High-Frequency vs. Theta-Burst TMS for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krajská zdravotní, a.s. - Nemocnice Most, o.z. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS-RCT-KZCR
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Major Depression
Keywords: TMS; iTBS; Transcranial magnetic stimulation; Theta burst stimulation; depression; anxiety; RCT
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study used a double-blind design. Participants were randomly assigned to receive either high-frequency rTMS or intermittent theta-burst stimulation but were not told which protocol they received. Clinical evaluators and most research staff involved in assessments were also blinded to treatment allocation. Only the technicians administering stimulation knew the protocol, and they were not involved in outcome assessments. To maintain blinding, both groups were informed that they were receiving an established rTMS treatment, and clinical raters avoided discussing protocol details with participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HF-rTMS (Active Comparator): High-frequency rTMS was delivered to the left dorsolateral prefrontal cortex using the 5 cm rule to localize the target site. Stimulation intensity was set at 100% of the resting motor threshold, determined by visible motor-evoked potentials in the right abductor pollicis brevis muscle. Each session consisted of 1500 pulses at 10 Hz, organized into 10 trains of 15 seconds (150 pulses per train) with 50-second inter-train intervals. Total stimulation time per session was approximately 12.5 minutes. A figure-of-eight coil (70BFX-LQC, Deymed Diagnostics) connected to a DuoMagXT-100 stimulator was used, with the coil positioned at ~45° from the midline, handle pointing posterolaterally.
  Interventions: Device: High-frequency repetitive transcranial magnetic stimulation
- iTBS (Active Comparator): Intermittent theta-burst stimulation (iTBS) was delivered to the left dorsolateral prefrontal cortex using the 5 cm rule for target localization. Stimulation intensity was set at 100% of the resting motor threshold, determined by motor-evoked potentials in the right abductor pollicis brevis muscle. Each session consisted of 600 pulses delivered in bursts of three 50 Hz pulses repeated every 200 ms. Trains of 2 seconds were followed by 8-second inter-train intervals. Total stimulation time per session was approximately 3 minutes and 20 seconds. A figure-of-eight coil (70HF-LQC, Deymed Diagnostics) connected to a DuoMagXT-100 stimulator was used, with coil orientation ~45° from the midline, handle pointing posterolaterally.
  Interventions: Device: Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: High-frequency repetitive transcranial magnetic stimulation — High-frequency rTMS was delivered to the left dorsolateral prefrontal cortex using the 5 cm rule to localize the target site. Stimulation intensity was set at 100% of the resting motor threshold, determined by visible motor-evoked potentials in the right abductor pollicis brevis muscle. Each session consisted of 1500 pulses at 10 Hz, organized into 10 trains of 15 seconds (150 pulses per train) with 50-second inter-train intervals. Total stimulation time per session was approximately 12.5 minutes. A figure-of-eight coil (70BFX-LQC, Deymed Diagnostics) connected to a DuoMagXT-100 stimulator was used, with the coil positioned at ~45° from the midline, handle pointing posterolaterally.
  Arms: HF-rTMS
Device: Intermittent Theta Burst Stimulation — Intermittent theta-burst stimulation (iTBS) was delivered to the left dorsolateral prefrontal cortex using the 5 cm rule for target localization. Stimulation intensity was set at 100% of the resting motor threshold, determined by motor-evoked potentials in the right abductor pollicis brevis muscle. Each session consisted of 600 pulses delivered in bursts of three 50 Hz pulses repeated every 200 ms. Trains of 2 seconds were followed by 8-second inter-train intervals. Total stimulation time per session was approximately 3 minutes and 20 seconds. A figure-of-eight coil (70HF-LQC, Deymed Diagnostics) connected to a DuoMagXT-100 stimulator was used, with coil orientation ~45° from the midline, handle pointing posterolaterally.
  Arms: iTBS

SUMMARY:
The goal of this clinical trial was to learn if two different types of repetitive transcranial magnetic stimulation (rTMS) could help treat depression and anxiety in adults with major depressive disorder.

The main questions it aimed to answer were:

Did high-frequency rTMS and intermittent theta-burst stimulation (iTBS) both reduce depressive symptoms? Did one treatment lead to greater improvement in anxiety symptoms?

Researchers compared people receiving high-frequency rTMS to those receiving iTBS to see if one worked better for mood and anxiety symptoms.

Participants:

Were randomly assigned to one of the two treatment groups. Received 10 stimulation sessions over two weeks (five sessions per week). Completed questionnaires and interviews on depression, anxiety, and stress before treatment, after two weeks, and again six weeks later.

DETAILED DESCRIPTION:
This randomized, double-blind clinical trial evaluated two established repetitive transcranial magnetic stimulation (rTMS) protocols-high-frequency rTMS (HF-rTMS) and intermittent theta-burst stimulation (iTBS)-delivered in a shortened, two-week treatment schedule for adults with major depressive disorder (MDD). The purpose was to determine whether a condensed regimen could provide effective relief of depressive and anxiety symptoms while improving treatment feasibility.

Design and Intervention A total of 108 participants with a primary diagnosis of MDD were randomized in a 1:1 ratio to receive either HF-rTMS (10 Hz stimulation) or iTBS, both targeting the left dorsolateral prefrontal cortex (DLPFC). Treatments were administered over 10 sessions in two consecutive weeks (five sessions per week).

HF-rTMS protocol: 1500 pulses per session at 10 Hz, delivered in 10 trains of 15 seconds each with 50-second inter-train intervals. Total session time: approximately 12.5 minutes.

iTBS protocol: 600 pulses per session, delivered as bursts of three 50 Hz pulses repeated at 200 ms intervals, with 2-second trains and 8-second inter-train intervals. Total session time: approximately 3 minutes and 20 seconds.

Stimulation intensity for both protocols was set at 100% of the participant's individual resting motor threshold.

Blinding and Assessments The trial employed a double-blind design: participants, clinical evaluators, and most research staff were unaware of treatment allocation. Independent clinicians performed structured interviews and validated rating scales before treatment (baseline), after two weeks of treatment, and at six-week follow-up.

Outcomes and Rationale The primary outcomes were changes in depressive symptoms measured by the Hamilton Depression Rating Scale (HAMD) and the Zung Self-Rating Depression Scale (SDS), and changes in anxiety symptoms measured by the Hamilton Anxiety Rating Scale (HAMA) and the Beck Anxiety Inventory (BAI). Secondary outcomes included perceived stress and self-reported depressive symptomatology.

This study was motivated by clinical and logistical considerations: standard rTMS protocols often require 4-6 weeks of treatment, which can be burdensome for patients and health systems. Evidence suggests that much of the therapeutic response occurs within the first 10-15 sessions, raising the possibility that shorter regimens may capture the critical therapeutic window.

By directly comparing HF-rTMS and iTBS within a condensed protocol, this trial aimed to clarify their relative antidepressant and anxiolytic efficacy, evaluate the durability of short-course treatment, and inform optimized approaches to neuromodulation in depression.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 to 90 years.
* Current major depressive disorder (MDD) as the primary diagnosis, confirmed according to the International Classification of Diseases, 10th Revision (ICD-10).
* All participants had to be evaluated by a board-certified psychiatrist trained in rTMS to confirm eligibility.
* Ability and willingness to provide written informed consent prior to study participation.

Exclusion Criteria

* Presence of ferromagnetic or electronic implants in the head or neck (e.g., pacemakers, aneurysm clips, cochlear implants, deep brain stimulators).
* Known seizure disorders (such as epilepsy) or significantly increased risk of seizures.
* Other major neurological diseases or conditions that would interfere with safe rTMS administration.
* Active psychotic symptoms or a primary psychotic disorder.
* Acute manic episode or recent hospitalization for mania or other severe psychiatric instability.
* Ongoing electroconvulsive therapy (ECT) treatment.
* Medication changes made during the study.
* Inability to comply with the treatment schedule (e.g., attendance problems, logistical barriers).
* Any medical or psychiatric condition judged by the investigators to compromise safety or data integrity.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Zung Self-Rating Depression Scale (SDS) | From baseline to post-treatment at 2 weeks and follow-up at 6 weeks.
  A 20-item self-reported questionnaire measuring depressive symptoms. Each item is scored 1-4, yielding a total raw score range of 20-80. Standardized scores are calculated by multiplying the raw score by 1.25, with higher scores reflecting greater severity of depression (≥50 = clinically significant depression).
Hamilton Depression Rating Scale (HAMD) | From baseline (before treatment) to post-treatment at 2 weeks and follow-up at 6 weeks.
  A structured interview conducted by a trained clinician to assess severity of depressive symptoms. The HAMD contains 17-21 items scored from 0 (absent) to 2 or 4 (severe), depending on the item. The total score ranges from 0 to 52, with higher scores indicating more severe depression. Common interpretation: 0-7 = normal, 8-16 = mild depression, 17-23 = moderate, ≥24 = severe.
Beck Anxiety Inventory (BAI) | From baseline to post-treatment at 2 weeks and follow-up at 6 weeks.
  A 21-item self-reported questionnaire assessing common symptoms of anxiety. Each item is rated 0 (not at all) to 3 (severe), with a total score range of 0 to 63. Higher scores indicate more severe anxiety (0-7 = minimal, 8-15 = mild, 16-25 = moderate, 26-63 = severe).
Hamilton Anxiety Rating Scale (HAMA) | From baseline to post-treatment at 2 weeks and follow-up at 6 weeks.
  A clinician-rated scale that assesses severity of anxiety symptoms. It has 14 items, each rated from 0 (not present) to 4 (severe). The total score ranges from 0 to 56, with higher scores indicating greater anxiety (≤17 = mild, 18-24 = moderate, 25-30 = severe). Includes subscores for psychological and somatic anxiety.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR-16) | From baseline to post-treatment at 2 weeks and follow-up at 6 weeks.
  A 16-item self-report scale assessing core symptoms of depression such as mood, sleep, appetite, and concentration. Each item is scored 0-3, with total scores ranging from 0 to 27. Higher scores represent greater severity (1-5 = mild, 6-10 = moderate, 11-15 = moderately severe, 16-20 = severe, ≥21 = very severe).
Perceived Stress Scale (PSS) | From baseline to post-treatment at 2 weeks and follow-up at 6 weeks.
  A 10-item self-report questionnaire measuring the degree to which participants perceive life situations as stressful. Each item is rated 0 (never) to 4 (very often), with total scores ranging from 0 to 40. Higher scores reflect higher perceived stress (0-13 = low, 14-26 = moderate, 27-40 = high stress).

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Albrecht, MD, Ph.D., Principal Investigator — Department of Psychiatry, Most Hospital, Krajská zdravotní a.s., Most, Czech Republic
Locations (1):
- Krajská zdravotní, a.s. - Nemocnice Most, o.z., Most, Ústecký kraj, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The main reasons are protection of participant privacy and confidentiality, as well as limitations in the consent form that did not include permission for public data sharing. Aggregate results are available in the published manuscript and can be provided upon reasonable request to the corresponding author.